CLINICAL TRIAL: NCT03326479
Title: Caris Molecular Intelligence® and Caris Centers of Excellence for Precision Medicine NetworkTM Retrospective Outcomes-Associated Database
Brief Title: POA Retrospective Repository
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Caris Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: COE-002-1116
Record Dates: First submitted 2017-10-19; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Oncology; Solid Tumor, Adult
Keywords: Molecular Profiling; Biomarker Analysis; Outcomes Database
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective: Subject who have previously had MI Profiling performed prior to 11/11/2016 are eligible for this study. No drug intervention is required for this study.
  Interventions: Diagnostic Test: Caris Molecular Intelligence Profile

INTERVENTIONS:
Diagnostic Test: Caris Molecular Intelligence Profile — A comprehensive biomarker testing

SUMMARY:
This repository is a multi-center, outcomes study designed to retrospectively collect data on the demographics, presentation, diagnosis, treatment, cost of associated care, quality of life, and outcomes of subjects utilizing Caris Molecular Intelligence® (CMI) Services for the treatment of cancer. Prior to enrolling a subject, the subject's physician will have made the independent decision whether or not to utilize the drug associations provided by CMI and made clinical treatment choices as appropriate. Thus, data captured and reported provides a "real world" perspective on diagnosis, treatment, cost, and outcomes.

DETAILED DESCRIPTION:
This repository is a multi-center, outcomes study designed to retrospectively collect data on the demographics, presentation, diagnosis, treatment, cost of associated care, quality of life, and outcomes of subjects utilizing Caris Molecular Intelligence® (CMI) Services for the treatment of cancer. Prior to enrolling a subject, the subject's physician will have made the independent decision whether or not to utilize the drug associations provided by CMI and made clinical treatment choices as appropriate. Thus, data captured and reported provides a "real world" perspective on diagnosis, treatment, cost, and outcomes.

Patients who have had CMI testing prior to the initial IRB submission date of November 11, 2016 for the respective site would be eligible to have their treatment and treatment response data entered into the study Database. All entered data would be de-identified. The patient's CMI biomarker results and treatment response data will be coupled together in order to allow the investigation of research questions concerning biomarker status and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Subject' s age must be greater than or equal to 18 years and must have received CMI testing prior to the initial protocol IRB submission date of November 11, 2016.

Exclusion Criteria:

* Due to the complexity of state and federal requirements governing the participation of prisoners in research, prisoners-patients shall not be approached for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject's who have had CMI testing prior to 11/11/2016 at one of the participating POA sites.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-11-30 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Data Gathering | 5 years per patient
  Documentation of the frequency of specific clinical events in relation to diagnosis, treatments and outcomes provided

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas